## EFFECT OF PLACING THE ENDOTRACHEAL TUBE BEYOND CERVICAL C7 LEVEL IN ANTERIOR CERVICAL DECOMPRESSION AND FUSION SURGERY: AN OBSERVATIONAL STUDY ON ENDOTRACHEAL CUFF PRESSURE CHANGES

Dr. Liu Chian Yong MD (UKM), MMED Anaesthesiology (UKM)

Dr. Noor Afifah binti Said (Alexandria University, Egypt )

UNIVERSITI KEBANGSAAN MALAYSIA (UKM)
18th June 2024

## **FLOWCHART**



- Intubation and placement of endotracheal cuff beyond C7.
- Inflate the ETT cuff to 20 cmH<sub>2</sub>0 and check for equal breath sound.
- Visualisation of carina using flexible fibreoptic scope.
- Reconfirmation of ETT placement using image-intensifier.
- Continuous monitoring of ETCP by connecting pilot balloon to the pressure transducer



- Primary objectives: Monitoring of pressure variation every 15 min. and record these ETCP
  - 1. ETCP<sub>base</sub> which is the baseline pressure after neck extension
  - 2. ETCP<sub>before</sub> before retraction of neck tissues
  - 3. ETCP<sub>retract</sub> during retraction of neck tissues
  - 4. ETCP<sub>after</sub> after the removal of retractors
- Secondary objectives :
  - Assess sore throat, dysphagia, and hoarseness of voice in recovery,
     6 hours, and 24 hours after extubation.